CLINICAL TRIAL: NCT03028662
Title: New Therapeutic Strategies for the Treatment of Alcohol Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gabriel Rubio Valladolid, MD (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Gabriel Rubio Valladolid, MD, Psychiatrist, MD, PhD, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-00463
Record Dates: First submitted 2016-10-11; First posted 2017-01-23 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Alcoholism
Keywords: Alcohol Dependence; Brain Connectivity; Inhibition
MeSH Terms: conditions — Alcoholism; Inhibition, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Immediate exposure (Experimental): Exposure to video on alcohol (update phase) followed (10 minutes) by the task of approach-avoidance of alcohol (extinction phase) (Retrieval-Extinction Learning), during 4 days of training.
  Interventions: Behavioral: Retrieval-Extinction Learning
- Delayed exposure (Active Comparator): Exposure to a video of alcohol consumption (update phase) followed (6 hours) by the task of approach-avoidance of alcohol (extinction phase) (Retrieval-Extinction Learning), during 4 days of training.
  Interventions: Behavioral: Retrieval-Extinction Learning
- No exposure (Active Comparator): Exposure to a video of neutral situations (update phase) followed (10 minutes) by the task of approach-avoidance of alcohol (extinction phase) (Retrieval-Extinction Learning), during 4 days of training.
  Interventions: Behavioral: Retrieval-Extinction Learning

INTERVENTIONS:
Behavioral: Retrieval-Extinction Learning — The intervention consists of the accomplishment of the task of approach-avoidance of alcohol during 4 days of training. Subjects are instructed to respond with an approach movement (pulling a lever) to neutral images and to respond with avoidance movement (pushing the lever) to images of alcohol.

SUMMARY:
This is an experimental study in which the efficacy of three psychophysiological intervention modalities based on retrieval-extinction procedures is analyzed.

DETAILED DESCRIPTION:
Behavioral inhibition processes are a particularly relevant in relapses of patients with alcohol dependence. One of the current behavioral techniques to improve inhibitory abilities of these patients is the alcohol Approach Avoidance Task (AAT). However, this technique could be more efficient if patients, before training in this task, were exposed to a variety of alcohol-conditioned stimuli (retrieval) and take advantage of the window period of reconsolidation of these memories to carry out this task (extinction training). This project will attempt to show the pattern of brain connectivity underlying retrieval-extinction learning, its relationship with markers such as Brain-Derived Neurotrophic Factor (BDNF) and their usefulness to reduce relapses of individual with alcohol dependence. To carry out this study 115 patients with alcohol dependence who will be randomized into three groups: Group 1 (N = 35) where the extinction training is performed within the window period (10 minutes); Group 2 (N = 35) extinction will take place outside the time window (6 hours); Group 3 (N = 35), these subjects will be exposed to "non-retrieval" but with extinction-training within the window period. Changes in connectivity will be assessed with Electroencephalogram (EEG) at baseline and after 4 training sessions, using the HERMES platform. BDNF levels will be determined as peripheral markers of neurogenesis. These changes will be are correlated with relapses in the 12 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol-dependent patients who have been detoxified and abstinent take 10-14 days.

Exclusion Criteria:

* Patients who do not sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2016-01; Primary Completion 2020-09 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Difference between pattern of brain connectivity after training-extinction and basal level | 2 days
Number of relapses during 3 months after training-extinction | 3 months

SECONDARY OUTCOMES:
Difference between plasma levels of BDNF after training-extinction and basal level | 2 days
Difference between attentional bias toward alcohol after training-extinction and basal level | 2 days
Difference between behavioral inhibition after training-extinction and basal level | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Rubio Valladolid, Psychiatrist, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiers RW, Eberl C, Rinck M, Becker ES, Lindenmeyer J. Retraining automatic action tendencies changes alcoholic patients' approach bias for alcohol and improves treatment outcome. Psychol Sci. 2011 Apr;22(4):490-7. doi: 10.1177/0956797611400615. Epub 2011 Mar 9. PMID 21389338